CLINICAL TRIAL: NCT06455553
Title: Interpretability of the Quantra® Viscoelastic Test in Patients With Haematological Malignancies With Profound Thrombocytopenia Below 50 G/L. First Exploratory Sub-study of the Global VISCOTHEM Project to Evaluate the Performance of VISCOelastic Tests in Predicting Bleeding in Thrombocytopenic Patients With Malignant Hemopathy.
Brief Title: Interpretability of the Quantra® Viscoelastic Test in Patients With Haematological Malignancies With Profound Thrombocytopenia Below 50x10 G/L.
Acronym: VISCOTHEM-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 24-01
Record Dates: First submitted 2024-06-04; First posted 2024-06-12 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Hematologic Malignancies; Thrombopenia
MeSH Terms: conditions — Hematologic Neoplasms; Thrombocytopenia | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (additional blood sample) (Other)
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — A blood sample will be taken from all patients included in the study. This blood sampling is an added act of the study. It will be performed as soon as possible after inclusion in the study. The total volume of blood drawn will be 12.1 mL. The following analyses will be performed: Quantra®, Rotem®, blood count, platelets, immature platelet count, plasma prothrombin time, activated partial thromboplastin time, International Normalized Ratio, fibrinogen.

SUMMARY:
The goal of this single-center, non-controlled, non-randomized exploratory clinical trial is to evaluate the interpretability of viscoelastic tests (Quantra® and ROTEM® type) in relation to platelet levels measured in standard biology in patients with haematological malignancies, hospitalized in day hospitals or full hematology wards, presenting thrombocytopenia strictly below 50 G/L.

Participants will undergo an additional blood sample to standard care. The total volume of blood drawn will be 12.1 mL. The following analyses will be performed: Quantra®, Rotem®, blood count, platelets, immature platelet count, plasma prothrombin time, activated partial thromboplastin time, International Normalized Ratio, fibrinogen.

ELIGIBILITY:
Inclusion Criteria:

* Patient age > 18 years old ;
* Patients who have been informed of the study and have freely given their informed consent to participate in the study;
* Patients with hematologic malignancies, treated or untreated, at any stage of treatment;
* Patient with thrombocytopenia strictly below 50 G/L on a blood sample taken less than 72 hours ago;
* Patient hospitalized in day hospitalization or in full hematology hospitalization;
* Patient covered by a French social security scheme.

Exclusion Criteria:

* Patients treated with antiplatelet agents or anticoagulants in preventive or curative doses;
* Patient with a history of thrombopathy;
* Patient with a history of haemostasis pathology at risk of haemorrhage or thrombosis;
* Pregnant or breast-feeding patients;
* Patients under guardianship;
* Patients who do not understand French;
* Patients under court protection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-06-26 (Actual); Primary Completion 2024-12-06 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the correlation between Quantra® (Clot firmness) and conventional biology results in patients with hematologic malignancies with platelet counts strictly below 50 G/L. | At baseline, before platelet transfusion
  Correlation coefficient (r²) and its 95% confidence interval (IC95) between patients' platelet levels obtained by conventional biology and Clot firmness (CS) obtained with Quantra®.
Evaluate the correlation between Quantra® (Platelet contribution to clot) and conventional biology results in patients with hematologic malignancies with platelet counts strictly below 50 G/L. | At baseline, before platelet transfusion
  Correlation coefficient (r²) and its 95% confidence interval (IC95) between patients' platelet levels obtained by conventional biology and Platelet contribution to clot (PCS) obtained with Quantra®.

SECONDARY OUTCOMES:
Evaluate the correlation between ROTEM® results and conventional biology results in patients with hematologic malignancies with platelet counts strictly below 50 G/L. | At baseline, before platelet transfusion
  Correlation coefficients (r²) and its 95% confidence interval (IC95) between patients' platelet levels obtained in conventional biology and the following measurements obtained in ROTEM® :
  1. MCFextem
  2. MCFfibtem
  3. CTextem
  4. MCEplatelets With MCEplatelets = [(100 × MCFextem)/(100 - MCFextem)] - [(100 × MCFfibtem)/(100 - MCFfibtem)]
Evaluate the correlation between Quantra® or ROTEM® results and platelet levels in the subpopulations of interest: patients with 0 to 9 G/L, 10 to 19 G/L and 20 to 49 G/L platelets. | At baseline, before platelet transfusion
  Stratify correlation analyses and their r² coefficients (IC95) on thrombocytopenia depth into three groups:
  1. 0 to 9 G/L
  2. 10 to 19 G/L
  3. 20 to 49 G/L
To assess the correlation between Quantra® or ROTEM® results and platelet levels in the subpopulations of interest: patients with bleeding and patients without bleeding. | At baseline, before platelet transfusion
  Stratify correlation analyses and their r² coefficients (IC95) on the presence or absence of bleeding at inclusion.
Evaluate the correlation between Quantra® and ROTEM® results. | At baseline, before platelet transfusion
  Matrix of correlation coefficients (r²) and IC95 between Quantra® and ROTEM® values.
Describe changes in Quantra®, ROTEM® and other hemostasis parameters after platelet transfusion in thrombocytopenic patients transfused as part of routine care. | Immediately after platelet transfusion
  Quantitative evolution of Quantra® (CS and PCS), ROTEM® (MCFextem MCFfibtem, CTextem, MCEplatelets), plasma prothrombin time, activated partial thromboplastin time, International Normalized Ratio, fibrinogen, hemoglobinemia, hematocrit and platelet count, immature platelets, leukocytes, neutrophils before and 1 hour after platelet transfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Adrien CONTEJEAN, Principal Investigator — Annecy Genevois Hospital
Locations (1):
- Centre Hospitalier Annecy Genevois, Annecy, France

IPD SHARING:
Plan to Share IPD: No